CLINICAL TRIAL: NCT02177968
Title: Public Health Concerns of Elderly Fallers and Non-fallers in a Southeastern Community of Brazil
Brief Title: Public Health Concerns of Elderly Fallers and Non-fallers in a Community
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Luciana Paludetti Zubieta Traldi, Department Social Medicine's Master, University of Sao Paulo
Other Study IDs: HCRP9879/2011
Record Dates: First submitted 2014-06-23; First posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Accidental Falls; Aging
Keywords: fall; elderly; characteristics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Elderly fallers or non-fallers: characteristics of these groups
  Interventions: Other: descriptive analysis of characteristics

INTERVENTIONS:
Other: descriptive analysis of characteristics — comparison between elderly fallers and non-fallers

SUMMARY:
The purpose of this study is to identify the prevalence and the characterization of health of elderly fallers and non-fallers in the southeastern community of Brazil in the state of São Paulo.

DETAILED DESCRIPTION:
The population consisted of 638 elderly individuals enrolled and attended by the teams of the Family Health Strategy in the city of Araraquara, São Paulo state. The sample was selected in a systematic way, considering the order of micro-areas, 1-7, which 10% sampling error, 15% rate answer. To this, instruments were used based SABE Study, Health Wellbeing and Aging modified, and the International Physical Activity Questionnaire (IPAQ), short version.

ELIGIBILITY:
Inclusion Criteria:

* People aged 60 years and over

Exclusion Criteria:

* Vestibular alteration
* Postoperative requiring continuous home
* Low vision or complete blind
* Bedridden
* Empty house
* Subjects without registration at the health family unity

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Healthy, Well-being and Aging questionnaire | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Luciana PZ Traldi, research, Principal Investigator
Locations (1):
- Educação Permanente, Prefeitura Municipal de Araraquara, Araraquara, São Paulo, Brazil